CLINICAL TRIAL: NCT00967187
Title: A Phase II Multicenter, Open-label, Randomized, Parallel Group, Study of Bevirimat in HIV-1 Positive Patients to Evaluate the Safety, Efficacy, and Pharmacokinetics of MPC-4326 Administered as Monotherapy for 14 Days and as Part of an Optimized Background Regimen for up to 72 Weeks.
Brief Title: Safety and Efficacy Study of MPC-4326 for Treatment of Patients With HIV-1 Infection.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Myrexis Inc. (Industry)
Responsible Party: Andrew Beelen, M.D., Study Director, Myriad Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MPC-4326-204; BVM Study 204
Record Dates: First submitted 2009-08-25; First posted 2009-08-27 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2010-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — bevirimat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MPC-4326 200 mg BID X 14 Days (Experimental)
  Interventions: Drug: bevirimat dimeglumine
- MPC-4326 300 mg BID X 14 Days. (Experimental)
  Interventions: Drug: bevirimat dimeglumine

INTERVENTIONS:
Drug: bevirimat dimeglumine — Patients will be treated with MPC-4326 200mg monotherapy for 14 days. Once the Day 15 viral load results become available, patients, who achieve at least a 0.5 log10 reduction in viral load by Day 15 will have the option to continue on both MPC-4326 and an optimized background regimen (OBR) through Week 72.
  Arms: MPC-4326 200 mg BID X 14 Days
Drug: bevirimat dimeglumine — Patients will be treated with MPC-4326, 300 mg monotherapy for 14 days. Once the Day 15 viral load results become available patients who achieve at least a 0.5 log10 reduction in viral load by Day 15 will have the option to continue on both MPC-4326 and an optimized background regimen (OBR) through Week 72.
  Arms: MPC-4326 300 mg BID X 14 Days.

SUMMARY:
To evaluate the antiretroviral activity and safety of 200 mg BID and 300 mg BID doses of MPC-4326 administered as monotherapy for 14 days to HIV-1 positive patients. Patients with an initial treatment response will have the option to continue MPC-4326 in combination with an Optimized Backround Regimen for a maximum of 72 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age at the time of screening.
* Have HIV-1-infection.
* Have a CD4+-lymphocyte count≥100 cells/mm3
* Have a screening plasma HIV-1 RNA value, measured by the Roche Amplicor assay, of 2,000 - 500,000 copies/mL (inclusive).
* Be free from any acute infection or serious medical illness within 14 days prior to study entry.

Exclusion Criteria:

* Current opportunistic infection characteristic of AIDS (Category C according to the CDC Classification System for HIV-1 Infection, 1993 Revised Version, Appendix A) that is diagnosed within 30 days or is poorly controlled.
* Patients with systolic blood pressure < 90 mmHg or > 140 mmHg or diastolic blood pressure < 60 mmHg or > 90 mmHg.
* A history of seizures (excluding pediatric febrile seizures) or current administration of prophylactic anti-seizure medications.
* A history of cerebrovascular accident (CVA) or transient ischemic attacks (TIA).
* Patients with the following laboratory parameters within 30 days prior to first dose of study drug: Hemoglobin < 10.0 g/dL for men and < 9.0 g/dL for women Neutrophil count < 1000/mm3 Platelet count < 50,000/mm3 AST or ALT > 2.5 times the upper limit of normal (patients with a positive HBV surface antigen or HCV antibody test at screening must have AST and ALT no more than 1.5 times the upper limit of normal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change in HIV-1 viral load from baseline to day 15 | 15 days

SECONDARY OUTCOMES:
To evaluate safety and tolerability | 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Beelen, MD, Study Director — Myrexis Inc.
Locations (4):
- Australia (4):
  - AIDS Research Initiative, Darlinghurst, New South Wales
  - Holdsworth House Medical Practice, Darlinghurst, New South Wales
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Taylor Square Private Clinic, Darlinghurst, New South Wales